CLINICAL TRIAL: NCT02569931
Title: Surgery for Patellofemoral Instability, is There Normal Gait
Brief Title: The Unstable Kneecap - the Impact of Anatomy on Function
Acronym: SPRING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15.0068; 15/SC/0512 (Other: REC/IRB reference)
Record Dates: First submitted 2015-09-30; First posted 2015-10-07 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2020-03

CONDITIONS: Patellar Dislocation
MeSH Terms: conditions — Patellar Dislocation | interventions — Gait Analysis; Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (Experimental): 36 participants recruited aged between 18 to 50 years of age
  Participants will be considered eligible for the study group if they have had two or more episodes of patellar dislocation or multiple episodes of subluxation with at least one of the following:
  i. Positive patellar apprehension test ii. Tenderness along the medial retinaculum iii. Abnormal patellar tracking or position.
  The study group will undergo gait analysis and electromyography before surgery and 6 months after surgery.
  During surgery the study group will undergo intra-operative tracking and pressure measurements.
  Interventions: Other: Gait analysis; Other: Electromyography; Procedure: Intra-operative tracking and pressure measurements
- control group (Other): 36 participants recruited aged between 18 to 50 years of age, matched for age and gender with the study group. Control participants should be healthy subjects with no history of knee injury or surgery.
  The control group will undergo gait analysis and electromyography.
  Interventions: Other: Gait analysis; Other: Electromyography

INTERVENTIONS:
Other: Gait analysis — Participants will be asked to walk on an instrumented treadmill. The study group will undergo gait analysis before surgery and 6 months after surgery. The control group will undergo gait analysis at one visit only.
Other: Electromyography — Participants in the study group will undergo electromyography before and 6 months after surgery. Participants in the control group will undergo electromyography at one visit only
  Other Names: muscle recording
Procedure: Intra-operative tracking and pressure measurements — Participants in the study group will undergo intra-operative tracking and pressure measurements to see if corrective surgery to stabilise the patella improves tracking and pressure measurements
  Arms: study group

SUMMARY:
The principal objective of the study is to find out which everyday activities make the kneecap unstable in people with patellofemoral instability.

Analysing how a patient with an unstable kneecap walks will help us to determine if surgery is successful in these patients by seeing if better scores on patient questionnaires are found in patients following surgery and whether these patients also have a better pattern of walking.

The investigators aim to use cameras and pressure pads to see how patients walk before and after surgery and see how this compares to patient scores on the questionnaires.

If the investigators find that patients walk better after surgery they can justify that surgery is worthwhile for the patient and cost effective for the NHS.

DETAILED DESCRIPTION:
Recruitment strategy:

Patients referred to a specialist patellofemoral clinic with an unstable kneecap(s) will be approached by the student and asked whether they would be interested in participating in the study (study group). Participants will be considered eligible for the study group if they have had two or more episodes of kneecap dislocation or many episodes of instability with at least one of the following: a feeling that the kneecap will dislocate with pressure, tenderness along the inner side of the knee and/or abnormal movement or position of the kneecap.

They will be given a Patient Information Sheet (PIS) and be given time during the clinic to ask questions about the study. During this first appointment as per routine current clinical practice they will have an X-ray of their knee and fill in standard questionnaires to score their knee function and pain (Norwich Patellofemoral Instability score, Kujala score, PainDetect score, catastrophising score). The patient's knees will also be examined by the consultant and a record made of the clinical findings. As per routine practice, a magnetic resonance imaging (MRI) scan of both knees will be organised for 4 weeks after the original appointment and measurements of knee shape recorded. A total of 32 patients will be invited to join the study to assess the movement of the kneecap in patients with kneecap instability.

A group of normal knees (control group) will be studied to compare the findings from students aged 18 to 50 years at St George's University of London allowing both age and gender to be matched to the study group . Students with no previous history of knee problems will be eligible to join the control group.

Inclusion criteria for both groups includes age 18-50 years, English language speakers, able to use public transport or drive.

Exclusion criteria for both groups includes pregnancy, breast feeding, inability to give informed consent, inflammatory arthropathy, osteoarthritis.

All participants in both the study and control groups will be provided with a Participant Information Sheet (PIS) outlining the study design, objectives, procedures, data management and dissemination plans. Participants will have a minimum of seven days to consider their participation in this study.

If a participant expresses an interest in participating, and after time to read, consider and discuss the PIS in clinic, they will be provided with an appointment at the MSk Lab at Imperial College. At the start of the assessment the participant will be asked about their potential eligibility based on the pre-defined eligibility criteria and will be provided with a further opportunity to ask any questions about the study. If they are still interested in participating, the potential participant will be asked to complete three Consent Forms and they will be enrolled in the study.

Data Collection:

Each patient participant will complete a Norwich Patellar Instability (NPI) Score questionnaire, a Kujala Patellofemoral Disorders Score, a PainDetect score and a Catastrophising score which are validated questionnaires. Baseline data recorded prior to testing will include: presence of joint hypermobility syndrome (Beighton score), age, gender, duration of symptoms, frequency of kneecap dislocation, knee range of motion, MRC (Medical Research Council) muscle strength (flexion and extension), previous patellofemoral joint surgery, family history of patellar instability and whether patellar instability is unilateral or bilateral. Basic demographic data for multi-variate regression analysis (e.g. Body Mass Index data) will also be collected, along with measurements such as leg length / height required for Hof scaling.

Testing Procedure:

Both the control and study group will have gait analysis measurements performed as a baseline for data collection. After a six minute acclimatization period at 4km/h on the instrumented treadmill (Kistler Gaitway, Kistler Instrument Corporation, Amherst, NY), the speed is increased until either the subject feels uncomfortable, or the walking performance deteriorates. The procedure generally takes 12 minutes of continuous walking. Following the flat ground assessment, the inclination is then increased in 5° increments at a steady 4 km/h, until either the subject feels uncomfortable, or the walking deteriorates. The treadmill is then ramped to an inclination of 7° downhill. The subject is then asked to walk initially at the same 4 km/h, and then at 0.5 km/h increments until they either feel uncomfortable, or the walking performance deteriorates.

At all incremental intervals of speed and inclination, data on the way participants walk are collected for both limbs with a by special plates under the treadmill track. Body weight scaling for leg length are also applied to the outputted mechanical data to correct for differences. All data are subject to averaging and filtering to handle the large amount of continuous data the machine captures, normally entailing a minimum of six steps for each limb.

The subject will be asked to reproduce activities that have been associated with subjective instability (e.g. running sideways, hopping, jumping, turning to look over a shoulder ) to determine if the subjective feeling of instability correlates with physiological changes in measurements captured on the instrumented treadmill. Electrical sensors on the skin will be used to detect muscle activity.

For the study group during corrective surgery to deepen the groove, special markers and three dimensional scanning will allow recording of kneecap movement without disturbing underlying tissues to see if there is a statistically significant measurable difference, and if this correlates to the change in performance/symptom scores.

Six months after surgery for the study group, gait analysis will be repeated at the MSk Lab as previously outlined to determine the effect of surgery. The patients will be asked again at this stage to fill in a Kujala and NPI score. It is anticipated that study subjects and controls will be recruited over six months with data collection finished by a year from enrolment of the first patient into the study.

Data Analysis:

The primary hypothesis of this study is that there will be a direct relationship between shape of the kneecap groove and participants' walking performance. This will be tested formally by comparing the measurements taken of the kneecap and groove shape, and those from the measurements of gait. The aim will be to see if surgery improves gait and stops the kneecap dislocating.

Study dissemination:

The findings of the study will be fed back to participants. Presentation of study findings will be made at a local level with submission of a presentation to a regional meeting and nationally prior to submission to journals offering open access publishing to allow dissemination to other professionals and the public.

ELIGIBILITY:
Inclusion Criteria:

* Patient subjects will be considered eligible for the study group if they have had two or more episodes of patellar dislocation or multiple episodes of subluxation with at least one of the following:

  * Positive patellar apprehension test
  * Tenderness along the medial retinaculum
  * Abnormal patellar tracking or position
* Control participants should be healthy subjects with no history of knee injury or surgery
* All participants will need to have the capacity to give informed consent in English
* All participants must be able to use public transport or drive

Exclusion Criteria:

* Pregnancy
* Breast feeding
* Arthritis
* Participation in other studies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal gait who have patellar instability | Before surgery
  Graphical measurement of raw kinematic data to include joint moments at ankle, knee and hip comparing patients with patellar instability to normal controls

SECONDARY OUTCOMES:
Number of patients with normal gait 6 months after surgery to correct patellar instability | 6 months
  Graphical measurement of raw kinematic data to include joint moments at ankle, knee and hip comparing patients after surgery to correct patellar instability to normal controls
Number of patients with normal ground reaction force 6 months after surgery to correct patellar instability | 6 months
  Measurement of ground reaction force of patients after surgery to correct patellar instability compared to normal controls
Number of patients with a change in patellar tracking at the time of surgery to correct patellar instability | during surgery
  Graphical presentation of patellar movement in three dimensions measured intra-operatively during corrective surgery
Number of patients with a change in patellar pressure at the time of surgery to correct patellar instability | during surgery
  Graphical presentation of patellar pressure in three dimensions measured intra-operatively during corrective surgery
Number of patients who have an abnormal EMG compared to normal controls | before surgery
  Electromyographic (EMG) output in graphical form comparing patients with patellar instability to normal controls
Number of patients with a change in EMG 6 months after surgery to correct patellar instability | 6 months
  Electromyographic (EMG) output in graphical form comparing patients before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Hing, FRCS, Study Chair — St George's, University of London
Locations (2):
- United Kingdom (2):
  - St George's Hospital, London
  - Imperial College London, London